CLINICAL TRIAL: NCT01410617
Title: The Effect of Prophylactic Hemodialysis on the Morbidity and Mortality of the Patients With Chronic Kidney Disease Stages 3-4 Undergoing Coronary Artery Graft Bypass
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Khomeini Hospital (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Reza Khatami, Member of research board of Nephrology ResearchCenter of Tehran University of Medical Sciences, Imam Khomeini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THC-473
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Kidney Disease stage3; Chronic Kidney Disease stage4; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Renal Dialysis

ARMS (2):
- dialysis (Active Comparator): the patients who undergo 3 sessions prophylactic hemodialysis
  Interventions: Procedure: hemodialysis
- control group (No Intervention): the patients who do not undergo hemodialysis

INTERVENTIONS:
Procedure: hemodialysis — 3 sessions hemodialysis before CABG
  Arms: dialysis

SUMMARY:
Coronary artery disease is a major cause of death in patients with renal dysfunction Among patients who undergo coronary artery bypass grafting ,renal dysfunction is known To be a major predictor of in-hospital and remote mortality As little is known about the impact of non-dialysis-dependent renal dysfunction on short and mid term Outcomes following coronary surgery we have decided to investigate the effect of prophylactic Hemodialysis on the mortality and morbidity of the patients with ckd (stage 3,4 ) and compare these Effect with the control group

ELIGIBILITY:
Inclusion Criteria:

* 80<age>18
* ckd patients with stage 3,4
* CABG for the first time

Exclusion Criteria:

* age<18
* previous CABG (coronary artery bypass grafting)
* AKI(acute kidney injury)
* dialysis patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
morbidity | the morbidity during the time of hospitalization until discharge (baseline) and six month later
  morbidity is defined as length of hospitalization,infection rate,duration of mechanical ventilation,bleeding complications,

SECONDARY OUTCOMES:
mortality | from the time of CABG (baseline) until six months later

CONTACTS AND LOCATIONS:
Overall Officials: Roghieh Borji, MD, Principal Investigator — Imam Khomeini Hospital; Mohammad R Khatami, MD, Study Director — Nephrology research Center; Seyyed Hossein Ahmadi, MD, Study Chair — Tehran Herat Center; Khosro Barkhordari, MD, Principal Investigator — Tehran Heart Center; Mohammad R Abbasi, MD, Principal Investigator — Nephrology Researc Center
Locations (1):
- Tehran Herat Center, Tehran, Tehran Province, Iran